CLINICAL TRIAL: NCT02084316
Title: Testing and Linkage to HIV Care in China: A Clustered Randomized Trial
Brief Title: Testing and Linkage to HIV Care in China
Acronym: CTN 0056
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Walter Ling, Professor and Founding Director Integrated Substance Abuse Programs, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA CTN 0056; U10DA013045 (NIH)
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-01

CONDITIONS: HIV
Keywords: China CDC; One4All testing algorithm; Guangxi Autonomous Region; Testing and Linkage to HIV Care in China
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One4All (Experimental): Participants with HIV-positive screening results on EIA will immediately have their blood drawn for CD4 and VL tests. Participants will receive post-screening test counseling. Two venous blood samples will be collected-one for immediate numeration of CD4 T-lymphocytes in the same hospital lave using PIMA POC CD4 analyzer and the other for later VL testing at the province CDC which takes 10-15 days. Participant will be notified in person of their CD4 results on the same day and provided post-CD4 test counseling. Counseling in the One4all intervention has been modified from the national SOC guidelines due to the different order of tests and the shortened time period between screening and CD4 testing. The participant will be provided with a tentative assessment of ART eligibility based on CD4 results and other factors. Those who are eligible for ART are encouraged to seek HIV care at the study hospitals via China's National Free ART program.
  Interventions: Behavioral: One4All
- Standard of Care (Active Comparator): The control condition is the current standard of care (SOC) utilized within the county hospitals in Guangxi China. This SOC has some variability between counties but in general follows the national policies. After the initial positive screening on EIA and subsequent repeat screening, participants will receive post-screening test counseling. Participants will then be tested by WB either at the same visit or a subsequent visit. The WB is sent offsite.
  After WB test results are reported to the hospital, the health care provider will contact the participant by phone. The participant will be asked to return to the hospital for results and post-WB test counseling. At this visit, a blood sample will be collected for CD4 testing, and an initial epidemiological investigation will be carried out.
  Once CD4 test results are available, participants must be located again to inform them of their results and ART eligibility and to provide post-CD4 test counseling.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: One4All — Participants with HIV-positive screening results on EIA will immediately have their blood drawn for CD4 and VL tests. Participants will receive post-screening test counseling. Two venous blood samples will be collected-one for immediate numeration of CD4 T-lymphocytes in the same hospital lave using PIMA POC CD4 analyzer and the other for later VL testing at the province CDC which takes 10-15 days. Participant will be notified in person of their CD4 results on the same day and provided post-CD4 test counseling. Counseling in the One4all intervention has been modified from the national SOC guidelines due to the different order of tests and the shortened time period between screening and CD4 testing. The participant will be provided with a tentative assessment of ART eligibility based on CD4 results and other factors. Those who are eligible for ART are encouraged to seek HIV care at the study hospitals via China's National Free ART program.
  Arms: One4All
Behavioral: Standard of Care — The control condition is the current standard of care (SOC) utilized within the county hospitals in Guangxi China. This SOC has some variability between counties but in general follows the national policies. After the initial positive screening on EIA and subsequent repeat screening, participants will receive post-screening test counseling. Participants will then be tested by WB either at the same visit or a subsequent visit. The WB is sent offsite.
  After WB test results are reported to the hospital, the health care provider will contact the participant by phone. The participant will be asked to return to the hospital for results and post-WB test counseling. At this visit, a blood sample will be collected for CD4 testing, and an initial epidemiological investigation will be carried out.
  Once CD4 test results are available, participants must be located again to inform them of their results and ART eligibility and to provide post-CD4 test counseling.
  Arms: Standard of Care

SUMMARY:
This study will evaluate the effects of a comprehensive approach (One4All) to increase the percentage of patients that receive their HIV testing results and counseling.

Primary Hypothesis: The One4All approach will increase the proportion of individuals who have completed all tests to confirm HIV diagnosis and received counseling within 30 days of screening HIV+, given they have screened HIV+ on the initial test, from 40% to 60%.

DETAILED DESCRIPTION:
The study consists of a cluster randomized trial (CRT) at county hospitals in Guangxi, China to assess the effectiveness of a structural intervention: a new testing algorithm, consisting of rapid point-of-care (POC) HIV and CD4 testing, with viral load (VL) testing in parallel, designed to ensure completeness of diagnostic assessment and accelerate time to ART initiation for patients deemed ART eligible (hereafter called the One4all Test Intervention).

This CRT will be conducted in 12 county general hospitals with an estimated average of 30 participants per hospital, totaling an estimated 360 participants. The unit of randomization is the hospital. Hospitals will be randomized to 1) theOne4all Test Intervention, or 2) the control condition, consisting of the current standard of care (SOC). The efficacy of the intervention will be evaluated at 1, 3, and 12 month follow-up assessments, and the differential efficacy for drug users (DUs) and non-drug users will be examined.

The study population will consist of adult participants who screen positive on an initial HIV enzyme immunoassay (EIA) in the 12 study hospitals. Since the study will be conducted in China, the vast majority of participants will be of Chinese or Asian descent. Women will be included and are expected to represent approximately 26% of the study population.

Eligibility Criteria:

Site Eligibility Criteria: The location of our study is Guangxi Zhuang Autonomous Region (Guangxi). We will select county-level general hospitals in order to ensure sufficient caseload at each hospital and homogeneity across hospitals. Guangxi counties usually have one general hospital (a limited number of counties have two or more general hospitals); this hospital has been designated as the only setting for delivering ART services in the respective county.

Study hospitals (n=12) will be selected based on the number of reported HIV positive screenings in the first 6 months of the previous year (2012) and on homogeneity in testing procedures between hospitals. Selected hospitals will have reported at least 30 patients who screened positive during the period of January to June 2012. Should more than 12 hospitals be identified the lowest screen positive hospital will not be considered for participation.

Participant Eligibility Criteria: Inclusion criteria will be 1) age 18 or older, 2) seeking care in study hospitals, 3) local residency or intent to live in study area for at least 90 days, and 4) received HIV positive results on the initial screening test. Any patient who does not meet these inclusion criteria will be excluded from the study. Additionally, patients who are pregnant or who have previously received confirmation of HIV infection in other care settings (e.g. CDC clinic, infectious disease hospital, sub-county-level hospital) are not eligible to participate. Any patient who is a prisoner or detainee at the time of initial screening will be excluded from the study. In the event that a participant is enrolled at a study hospital and subsequently incarcerated, data will be collected.

ELIGIBILITY:
Inclusion Criteria:

Participating individuals must:

1. Be at least 18 years old
2. Be an inpatient or outpatient seeking care in study hospitals
3. Test positive on an initial EIA HIV screen
4. Have local residency or intent to live in study area for at least 90 days

Exclusion Criteria:

Individuals will be excluded from study participation if they:

1. Do not meet any one or more of the above inclusion criteria
2. Test result negative on initial EIA HIV screen
3. Have previously received confirmation on HIV infection in the study hospital or in any other setting (e.g., CDC clinic, infectious disease hospital, sub-county-level hospital)
4. Are prisoners or detainees at the time of initial screening
5. Are pregnant women (pregnant women are subject to mandatory testing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Receipt of post-test results and counseling following testing completeness | 30 days
  The numerator is the number of HIV-positive participants who have received post-test results and counseling within 30 days of initial screening blood draw. The denominator is the number of participants who screened positive on the initial HIV EIA in the study arm (control or intervention).

SECONDARY OUTCOMES:
Proportion of treatment-eligible participants with CD4 < 350 | 90 days
  A secondary outcome is the proportion of treatment-eligible participants with CD4< 350 cells/mm3 who have initiated ART within 90 days of an initial positive HIV screening. We will define the secondary endpoint variable for hypothesis as a binary variable. If a participant with CD4 <350 cells/mm3 initiates ART within 90 days of a positive screening, the variable is defined equal to one. Otherwise, the variable is defined equal to zero. All participants who screened HIV-positive on the initial EIA at screening will be included in the analysis.

OTHER OUTCOMES:
Proportion of participants who have viral suppression based on the 12-month viral load test. | 12 months
  A tertiary outcome is the proportion of participants who have viral suppression based on the 12-month viral load test, where viral suppression is defined as viral load < 200 copies/mL We will define the tertiary endpoint variable as a binary variable. If a participant with VL < 200 copies/mL at 12 months after initial screening, the variable is defined equal to one. Otherwise, the variable is defined equal to zero. All participants who screened HIV-positive on the initial EIA at screening will be included in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Zunyou Wu, MD, PhD, Principal Investigator — National Center for AIDS/STD Control and Prevention; Walter Ling, MD, Principal Investigator — University of California, Los Angeles; Roger Detels, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (12):
- China (12):
  - Fusui County People's Hospital, Chongzuo, Guangxi
  - Ningming County People's Hospital, Chongzuo, Guangxi
  - Daxin County People's Hospital, Chongzu, Guangxi
  - Lingui County People's Hospital, Guilin, Guangxi
  - Lipu County People's Hospital, Guilin, Guangxi
  - Duan County People's Hospital, Hechi, Guangxi
  - Xiangzhou County People's Hospital, Laibin, Guangxi
  - Rongan County People's Hospital, Liuchow, Guangxi
  - Longan County People's Hospital, Nanning, Guangxi
  - Lingshan County People's Hospital, Qingzhoucun, Guangxi
  - Cenxi County People's Hospital, Wuzhou, Guangxi
  - Bobai County People's Hospital, Yulin, Guangxi

REFERENCES:
- [Derived] Wu Z, Tang Z, Mao Y, Van Veldhuisen P, Ling W, Liu D, Shen Z, Detels R, Lan G, Erinoff L, Lindblad R, Gu D, Tang H, Hu L, Zhu Q, Lu L, Oden N, Hasson AL, Zhao Y, McGoogan JM, Ge X, Zhang N, Rou K, Zhu J, Wei H, Shi CX, Jin X, Li J, Montaner JSG. Testing and linkage to HIV care in China: a cluster-randomised trial. Lancet HIV. 2017 Dec;4(12):e555-e565. doi: 10.1016/S2352-3018(17)30131-5. Epub 2017 Aug 31. PMID 28867267
- [Derived] Mao Y, Wu Z, McGoogan JM, Liu D, Gu D, Erinoff L, Ling W, VanVeldhuisen P, Detels R, Hasson AL, Lindblad R, Montaner JSG, Tang Z, Zhao Y. Care cascade structural intervention versus standard of care in the diagnosis and treatment of HIV in China: a cluster-randomized controlled trial protocol. BMC Health Serv Res. 2017 Jun 12;17(1):397. doi: 10.1186/s12913-017-2323-z. PMID 28606085
- Available data/document: Study Protocol: CTN0056 — http://ctndisseminationlibrary.org/protocols/ctn0056.htm